CLINICAL TRIAL: NCT05335915
Title: Acute Pharmacokinetic and Pharmacodynamic Effects of "Tobacco-Free" Oral Nicotine Pouches in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00318560; 1R01DA055962-01 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Nicotine Withdrawal; Nicotine Addiction; Drug Effect
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Tobacco Products

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Care Provider
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Original/Tobacco Flavored Pouch (low nicotine dose) (Experimental): participants will use a tobacco flavored pouch (4mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Original/Tobacco Flavored Pouch (high nicotine dose) (Experimental): participants will use a tobacco flavored pouch (8mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Mint/Menthol Flavored Pouch (low nicotine dose) (Experimental): participants will use a mint/menthol flavored pouch (4mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Mint/Menthol Flavored Pouch (high nicotine dose) (Experimental): participants will use a mint/menthol flavored pouch (8mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Fruit Flavored Pouch (low nicotine dose) (Experimental): participants will use a fruit flavored pouch (4mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Fruit Flavored Pouch (high nicotine dose) (Experimental): participants will use a fruit flavored pouch (8mg nicotine dose)under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Nicotine
- Own brand cigarettes (Active Comparator): participants will smoke participants' own brand of cigarettes under both controlled (experimenter-directed) and ad libitum use conditions
  Interventions: Other: Cigarette

INTERVENTIONS:
Other: Nicotine — Nicotine pouches will be self-administered
  Other Names: Tobacco
  Arms: Fruit Flavored Pouch (high nicotine dose); Fruit Flavored Pouch (low nicotine dose); Mint/Menthol Flavored Pouch (high nicotine dose); Mint/Menthol Flavored Pouch (low nicotine dose); Original/Tobacco Flavored Pouch (high nicotine dose); Original/Tobacco Flavored Pouch (low nicotine dose)
Other: Cigarette — Cigarette will be smoked
  Other Names: Nicotine; Tobacco
  Arms: Own brand cigarettes

SUMMARY:
The purpose of the present study is to examine the pharmacokinetics and pharmacodynamics of "tobacco-free" oral nicotine pouches, at various doses and flavors, in healthy adult smokers. The study will utilize a within-subjects, double-blind design. Upon enrollment, participants will complete 7 dosing conditions: tobacco-flavored pouch (low or high nicotine dose), mint/menthol-flavored pouch (low or high nicotine dose), and fruit-flavored pouch (low or high nicotine dose); participants will also complete a condition where the participants will smoke participants' preferred brand of cigarettes. In each experimental session, participants will complete 2 product-use bouts. In bout 1, the participants will use a single product (pouch or cigarette) for a fixed period under controlled conditions. In bout 2, participants will be given 2 hours to use participants' assigned product ad libitum.

DETAILED DESCRIPTION:
The purpose of the present study is to examine the pharmacokinetics and pharmacodynamics of "tobacco-free" oral nicotine pouches, at various doses and flavors, in healthy adult smokers. The study will utilize a within-subjects, double-blind design. Upon enrollment, participants will complete 7 dosing conditions: tobacco-flavored pouch (low or high nicotine dose), mint/menthol-flavored pouch (low or high nicotine dose), and fruit-flavored pouch (low or high nicotine dose); participants will also complete a condition where the participants will smoke participants' preferred brand of cigarettes. In each experimental session, participants will complete 2 product-use bouts. In bout 1, the participants will use a single product (pouch or cigarette) for a fixed period under controlled conditions. In bout 2, participants will be given 2 hours to use participants' assigned product ad libitum. Blood specimens will be obtained throughout the sessions to characterize the pharmacokinetics of nicotine and various pharmacodynamic outcomes (subjective drug effects, tobacco withdrawal symptoms, vital signs) will also be assessed. These procedures will be completed 7 separate times (on separate visits) by each participant (sessions will be separated by at least 48 hours).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 21 years old
2. good general health based on screening procedures (e.g., physical exam, blood testing)
3. vital signs in normal range (resting heart rate less than 100bpm, systolic blood pressure less than 150mmHg, diastolic blood pressure less than 90mmHg)
4. negative urine test for illicit drug use (excluding THC) and negative breath alcohol test at screening and before each session
5. self-report currently smoking daily
6. self-report at least a one year history of regular smoking
7. exhaled breath CO greater than or equal to 10ppm and urine cotinine greater than 100 ng/ml at screening
8. meet criteria for at least mild tobacco use disorder
9. no self-reported regular use of other tobacco products (e.g., smokeless products, e-cigarettes) in the past 30 days
10. no self-reported prior use of novel oral nicotine pouches
11. exhaled breath CO less than 10 ppm upon arrival for each study session.

Exclusion Criteria:

1. Psychoactive drug use (aside from cannabis, nicotine, alcohol, or caffeine) in past month
2. Current use of over-the-counter (OTC) drugs, supplements/vitamins, or prescription medications that, in the opinion of the investigators or medical staff, will impact safety
3. Use of cannabis >4 times per week
4. History of or current significant medical condition that, in the opinion of the investigators or medical staff, will impact safety
5. Current psychiatric condition or substance use disorder (aside from tobacco use disorder) that, in the opinion of the investigators or medical staff, will impact safety or study outcomes
6. Women who are pregnant, planning to become pregnant, or are breast-feeding
7. Currently seeking treatment to quit smoking or currently using a nicotine/tobacco cessation product.
8. Enrollment in another clinical trial in the past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of nicotine as assessed by the Cmax | Up to 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Maximum concentration (Cmax), is the highest plasma nicotine concentration reached during a session and provides important insight into the abuse liability of a tobacco product.
Pharmacokinetics of nicotine as assessed by the AUC | Up to 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Area under the curve (AUC), represents the total nicotine exposure during an entire session and provides important insight into the abuse liability of a tobacco product.
Subjective ratings of "Like Drug Effect" as assessed by the Drug Effect Questionnaire | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "like drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Subjective ratings of "Pleasant Drug Effect" as assessed by the Drug Effect Questionnaire | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "pleasant drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Subjective ratings of "take again" as assessed by the Drug Effect Questionnaire | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "take again". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Subjective ratings of "urge to smoke" as assessed by the Hughes-Hatsukami Withdrawal Questionnaire | 6.5 hours
  The HHWS will be used to obtain subjective ratings of "urge to smoke". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Subjective ratings of "craving to smoke" as assessed by the Hughes-Hatsukami Withdrawal Questionnaire | 6.5 hours
  The HHWS will be used to obtain subjective ratings of "craving to smoke". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

SECONDARY OUTCOMES:
Pharmacokinetics of nicotine as assessed by the Tmax | Up to 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Time to maximum concentration (Tmax), is the time (in minutes) to reach Cmax. This is another measure relevant for abuse liability.
Tobacco withdrawal symptoms as assessed by the Tiffany-Drobes QSU brief-Factor 1 | 6.5 hours
  The QSU-brief factor 1 (intention to smoke) measures tobacco withdrawal symptoms using 5 items; scores are summed to produce a single score ranging from 0 to 30
Tobacco withdrawal symptoms as assessed by the Tiffany-Drobes QSU brief-Factor 2 | 6.5 hours
  The QSU-brief factor 2 (anticipation of relief) measures tobacco withdrawal symptoms using 5 items; scores are summed to produce a single score ranging from 0 to 24
Topography as assessed by the total time of use | 2 hours
  During the 2 hour ad libitum bout, topography will be collected. The total time of use (out of 2 hours) will be assessed.
The Direct Effects of Nicotine Scale (DENS) | 6.5 hours
  The DENS will assess nicotine-specific effects. Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Perceived strength of effects as assessed by the Drug Effect Questionnaire | 6.5 hours
  The DEQ will assess subjective ratings for "feel drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Negative and aversive effects as assessed by the Drug Effect Questionnaire | 6.5 hours
  The DEQ will assess subjective ratings for "dislike drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No